CLINICAL TRIAL: NCT02387853
Title: Safety and Effect of LEO 90100 Aerosol Foam on the HPA Axis and Calcium Metabolism in Adolescent Subjects (Aged 12 to < 17 Years) With Plaque Psoriasis
Brief Title: Safety and Efficacy of Once Daily Topical Treatment With LEO 90100 Aerosol Foam in Adolescent Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0053-1108
Record Dates: First submitted 2015-03-12; First posted 2015-03-13 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LEO 90100 (Experimental)
  Interventions: Drug: LEO 90100

INTERVENTIONS:
Drug: LEO 90100

SUMMARY:
An international, multi-centre, prospective, open-label, non-controlled, single-group, 4-week trial in adolescent subjects with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria (all subjects)

* Psoriasis vulgaris on trunk and/or limbs affecting at least 2% BSA.
* Psoriasis vulgaris on the scalp affecting at least 10% of total scalp area.
* A total psoriatic involvement on trunk, limbs and scalp not exceeding 30% BSA.
* PGA score of at least mild on trunk and/or limbs at SV1, SV2 and V1.
* PGA score of at least mild on scalp at SV1, SV2 and V1.
* A serum albumin-corrected calcium below the upper reference limit at SV2.

Inclusion Criteria (for subjects performing HPA axis assessment)

* Psoriasis vulgaris on trunk and/or limbs affecting at least 10% BSA.
* Psoriasis vulgaris on the scalp affecting at least 20% of total scalp area.
* PGA score of at least moderate on trunk and limbs at SV1, SV2 and V1.
* PGA score of at least moderate on scalp at SV1, SV2 and V1.
* Normal HPA axis function at SV2 (serum cortisol concentration above 5 mcg/dl before ACTH challenge and serum cortisol concentration above 18 mcg/dl 30 minutes after ACTH challenge).

Exclusion Criteria (all subjects):

* A history of hypersensitivity to any component of LEO 90100.
* Systemic treatment with biological therapies (marketed or not marketed), with a possible effect on scalp and/or body psoriasis within the following time period prior to V1 and during the trial:

  1. etanercept - within 4 weeks prior to V1
  2. adalimumab, infliximab - within 2 months prior to V1
  3. ustekinumab - within 4 months prior to V1
  4. experimental products - within 4 weeks/5 half-lives (whichever is longer) prior to V1
* Systemic treatment with therapies other than biologicals, with a possible effect on scalp and/or body psoriasis (e.g. methotrexate, retinoids, immunosuppressants) within 4 weeks prior to V1 or during the trial.
* PUVA therapy within 4 weeks prior to V1.
* UVB therapy within 2 weeks prior to V1 or during the trial.

Exclusion Criteria (for subjects performing HPA axis assessment):

* A history of serious allergy, allergic asthma or serious allergic skin rash.
* Known or suspected hypersensitivity to any component of CORTROSYN® (including ACTH/cosyntropin/tetracosactide)
* Systemic treatment with corticosteroids (including inhaled and nasal steroids) within 12 weeks prior to SV2 or during the trial.
* Oestrogen therapy (including contraceptives) or any other medication known to affect cortisol levels or HPA axis integrity within 4 weeks prior to SV2 or during the trial.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Seyger, MD, Principal Investigator — UMC St Radboud
Locations (9):
- United States (6):
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Redwood Family Dermatology, Santa Rosa, California
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Greenwich Village Dermatology, New York, New York
  - Skin Speciality Dermatology, New York, New York
  - Dermatology Treatment and Research Center PA, Dallas, Texas
- UMC St Radboud, Nijmegen, Netherlands
- MULTIKLINIKA SALUTE Sp zo.o., Katowice, Poland
- Spitalul Clinic de Boli Infectioase si Tropicale, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 117 subjects were enrolled, this number includes all subjects who provided consent for participation in the trial and were screened. Out of the 117 subjects who were screened, 106 subjects met all inclusion criteria and none of the exclusion criteria, and were started on treatment in the LEO 90100 arm.
Groups:
- LEO 90100: LEO 90100, an aerosol foam formulation containing calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) was applied once daily to body and scalp psoriasis lesions.
Period: Overall Study
Arm/Group | LEO 90100
Started | 106
Completed | 103
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Of the 117 subjects who were enrolled in the trial and screened, 106 subjects met all inclusion criteria and none of the exclusion criteria. These 106 subjects comprise the Baseline Analysis Population.
Groups:
- LEO 90100: LEO 90100, an aerosol foam formulation containing calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) was applied once daily to body and scalp psoriasis lesions. This arm contains all 106 subjects that were assigned to treatment and constitutes the full analysis set and the safety analysis set. 33 subjects in this arm performed additional baseline and post-baseline HPA axis assessments and constitute the per protocol analysis set.
Arm/Group | LEO 90100
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 103
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 102
  Native Hawaiian or Other Pacific Islander | 1
  Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 9
  Romania | 32
  United States | 2
  Poland | 63
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is based on skin reaction to first 30-45 minutes sun exposure after a winter with no sun exposure:
  Type I: Unexposed skin color: white, always burns easily, never tans. Type II: Unexposed skin color: white, always burns easily, tans minimally. Type III: Unexposed skin color: white, burns moderately, tans gradually (light brown).
  Type IV: Unexposed skin color: white, burns minimally, always tans well (moderate brown).
  Type V: Unexposed skin color: brown, rarely burns, tans profusely (dark brown). Type VI: Unexposed skin color: black, never burns, deeply pigmented.
  Participants
    Type I | 5
    Type II | 44
    Type III | 46
    Type IV | 10
    Type V | 1
Height [Mean (Standard Deviation); unit: cm] | 165.79 (9.77)
Weight [Mean (Standard Deviation); unit: kg] | 60.01 (14.41)
Duration of plaque psoriasis [Mean (Standard Deviation); unit: years] | 4.3 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Number of subjects with adverse events in the safety analysis set, defined by excluding subjects from the full analysis set who either received no treatment with the IMP and/or for whom no post-baseline safety evaluations are available.
Time Frame: From Week -1 to Week 8
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 106
Participants
  Upper respiratory tract infection | 8
  Nasopharyngitis | 4
  Folliculitis | 1
  Impetigo | 1
  Oral herpes | 1
  Pharyngitis | 1
  Pulpitis dental | 1
  Rhinitis | 1
  Acne | 2
  Erythema | 1
  Pruritus generalised | 1
  Psoriasis | 1
  Skin reaction | 1
  Application site pain | 1
  Product physical consistency issue | 1
  Arthralgia | 1
  Myalgia | 1
  Myopia | 1
  Arthropod bite | 1
  Haemangioma of liver | 1
  Skin neoplasm excision | 1

2. Primary Outcome: Number of Subjects With Serum Cortisol Concentration of ≤18 mcg/dl at 30 Minutes After ACTH-challenge at Week 4
Description: Number of subjects with serum cortisol concentration of ≤18 mcg/dl at 30 minutes after ACTH-challenge at Week 4 in the per protocol analysis set, defined as all subjects from the full analysis set who were in the HPA axis cohort but excluding subjects who did not receive any treatment with the IMP, did not provide any results for the HPA axis test at Week 4, or did not meet the inclusion criterion concerning evidence of normal adrenal function at baseline.
Time Frame: 30 minutes after ACTH-challenge at Week 4
Population: Per protocol analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 33
Participants
  Serum cortisol equal to or below 18 mcg/dl | 3
  Serum cortisol above 18 mcg/dl | 30

3. Primary Outcome: Change in Albumin-corrected Serum Calcium From Baseline to Week 4
Description: Change in albumin-corrected serum calcium from baseline to Week 4 in safety analysis set. The safety analysis set, defined by excluding subjects from the full analysis set who either received no treatment with the IMP and/or for whom no post-baseline safety evaluations are available.
Time Frame: From baseline to Week 4
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | LEO 90100
Number analyzed (Participants) | 101
mmol/L | -0.016 (0.119)

4. Primary Outcome: Change in Calcium Excretion in 24-hour Urine From Baseline to Week 4
Description: Change in calcium excretion in 24-hour urine collection from baseline to Week 4 in the 24-hour urine HPA set, defined as all subjects in the safety analysis set. The safety analysis set is defined, according to the Consolidated Trial Protocol, by excluding subjects from the full analysis set who either received no treatment with the IMP and/or for whom no post-baseline safety evaluations are available.
Time Frame: From baseline to Week 4
Population: 24-hour urine HPA set
Measure: Mean (Standard Deviation); unit: mmol/24hr
Arm/Group | LEO 90100
Number analyzed (Participants) | 32
mmol/24hr | -0.335 (2.076)

5. Primary Outcome: Change in Calcium:Creatinine Ratio in 24-hour Urine From Baseline to Week 4
Description: Change in calcium:creatinine ratio in 24-hour urine collection from baseline to Week 4 in the 24-hour urine in HPA set, defined as all subjects in the safety analysis set who underwent HPA-axis testing.
Time Frame: From baseline to Week 4
Population: 24-hour urine in HPA set
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 90100
Number analyzed (Participants) | 31
mmol/g | -0.2892 (2.1185)

6. Secondary Outcome: Number of Subjects With Serum Cortisol Concentration ≤18 mcg/dL at Both 30 and 60 Minutes After ACTH-challenge at Week 4
Description: Number of subjects with serum cortisol concentration ≤18 mcg/dL at both 30 and 60 minutes after ACTH-challenge at Week 4 in the per protocol analysis set, defined as all subjects from the full analysis set who were in the HPA axis cohort but excluding subjects who did not receive any treatment with the IMP, did not provide any results for the HPA axis test at Week 4, or did not meet the inclusion criterion concerning evidence of normal adrenal function at baseline.
Time Frame: 30 and 60 minutes after ACTH-challenge at Week 4
Population: Per protocol analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 33
Participants
  Serum cortisol equal to or below 18 mcg/dL | 1
  Serum cortisol above 18 mcg/dl | 32

7. Secondary Outcome: Change in Calcium:Creatinine Ratio in Spot Urine Samples From Baseline to Week 4
Description: Change in calcium:creatinine ratio in spot urine samples from baseline to Week 4 in the spot urine non-HPA set, defined as all subjects in the safety analysis set who did not undergo HPA-axis testing.
Time Frame: From baseline to Week 4
Population: Spot urine non-HPA set
Measure: Mean (Standard Deviation); unit: mmol/g
Arm/Group | LEO 90100
Number analyzed (Participants) | 48
mmol/g | 0.4620 (1.8892)

8. Secondary Outcome: Number of Subjects With 'Treatment Success' According to Physician's Global Assessment (PGA) on Body
Description: Number of subjects with 'treatment success' according to Physician's Global Assessment (PGA) on Body in the full analysis set, defined as the 106 subjects assigned to treatment. Treatment success was defined as 'clear' or 'almost clear' for subjects with at least 'moderate' disease at baseline according to the PGA, and defined as 'clear' for subjects with mild disease at baseline according to the PGA.
Time Frame: Week 4
Population: Full analysis set. 3 subjects withdrew from the trial prior to the Week 4 visit, the remaining 103 subjects were included in the analysis of this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 103
Participants
  Yes | 74
  No | 29

9. Secondary Outcome: Number of Subjects With 'Treatment Success' According to Physician's Global Assessment (PGA) on Scalp
Description: Number of subjects with 'treatment success' according to Physician's Global Assessment (PGA) on Scalp in the full analysis set, defined as the 106 subjects assigned to treatment. Treatment success was defined as 'clear' or 'almost clear' for subjects with at least 'moderate' disease at baseline according to the PGA, and defined as 'clear' for subjects with mild disease at baseline according to the PGA.
Time Frame: Week 4
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 103
Participants
  Yes | 78
  No | 25

10. Secondary Outcome: Percentage Change in PASI From Baseline to Week 4
Description: Percentage change in Psoriasis area and severity index (PASI) score from baseline to Week 4. Psoriasis area and severity index (PASI) assesses extent and severity of clinical signs of psoriasis vulgaris. Body surface is divided in 4 ares: head (incl. neck), arms (incl. hands), trunk (incl. flexures) and legs (incl. buttocks and feet). Each area is scored from 0-6 for extent of psoriasis and from 0-4 for redness, thickness, and scaliness, and an area PASI score is calculated. The total PASI score is calculated from each area's score. The PASI score ranges from 0 (clear skin) to 72 (maximum disease), a PASI score higher than 10 generally corresponds to moderate-to-severe disease.
Time Frame: From baseline to Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage change in PASI
Arm/Group | LEO 90100
Number analyzed (Participants) | 103
Percentage change in PASI | -82.05 (17.87)

11. Secondary Outcome: Number of Subjects With 'Treatment Success' According to the Subject's Global Assessment of Disease Severity on the Body at Week 4
Description: Number of subjects with 'treatment success' according to the Subject's Global Assessment of disease severity on the body at Week 4 in the full analysis set, defined as the 106 subjects assigned to treatment. Treatment success was defined as 'clear' or 'very mild' according to the Subject's Global Assessment of disease severity.
Time Frame: Week 4
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 103
Participants
  Yes | 86
  No | 17

12. Secondary Outcome: Number of Subjects With 'Treatment Success' According to the Subject's Global Assessment of Disease Severity on the Scalp at Week 4
Description: Number of subjects with 'treatment success' according to the Subject's Global Assessment of disease severity on the scalp at Week 4 in the full analysis set, defined as the 106 subjects assigned to treatment. Treatment success was defined as 'clear' or 'very mild' according to the Subject's Global Assessment of disease severity.
Time Frame: Week 4
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 90100
Number analyzed (Participants) | 103
Participants
  Yes | 84
  No | 19

13. Secondary Outcome: Change in Itch as Assessed on a Visual Analog Scale (VAS) From Baseline to Week 4
Description: Change in itch as assessed on a visual analog scale (VAS) from baseline to Week 4 in the full analysis set, defined as the 106 subjects assigned to treatment. The assessments were made on a 100 mm (100 mm = 10 cm) horizontal VAS anchored at 0 ('no itch at all') and 10 ('worst itch you can imagine'). Subjects were asked to put a vertical line on the scale at the spot he/she felt best reflected the maximal itch intensity during the last 24 hours. The distance from 0 to the subject's indication line was measured in mm, thus higher scores indicated a worse outcome.
Time Frame: From baseline to Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm on VAS scale
Arm/Group | LEO 90100
Number analyzed (Participants) | 103
mm on VAS scale | -32.5 (27.3)

ADVERSE EVENTS:
Time Frame: From Day -28 up to Day 56
Description: During the trial, the investigator followed up all AEs (SAEs) until the final outcome was determined. After a subject had left the trial, the investigator followed up all non-serious AEs classified as possibly or probably related to the IMP for 14± 2 days or until the final outcome was determined, whichever came first. SAEs were followed up until a final outcome had been determined, that is, the follow-up could continue beyond the end of the trial.
Groups:
- LEO 90100: LEO 90100, an aerosol foam formulation containing calcipotriol 50 mcg/g (as hydrate) and betamethasone 0.5 mg/g (as dipropionate) was applied once daily to body and scalp psoriasis lesions. This arm contains all 106 subjects that were assigned to treatment and constitutes the full analysis set and the safety analysis set. 33 subjects in this arm performed additional HPA axis assessments and constitute the per protocol analysis set.
Arm/Group | LEO 90100
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 22/106
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 90100 (N=106)
Upper respiratory tract infection (Infections and infestations) | 8 (8)
Nasopharyngitis (Infections and infestations) | 4 (4)
Folliculitis (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Application site pain (General disorders) | 1 (1)
Product physical consistency issue (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myopia (Eye disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.

DOCUMENTS (2):
  • Study Protocol (2016-08-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT02387853/Prot_001.pdf
  • Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT02387853/SAP_000.pdf